CLINICAL TRIAL: NCT07095621
Title: Feasibility and Effectiveness of Three-day Discharge After Distal Pancreatectomy
Acronym: 3DD
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Nicolò Pecorelli, Surgeon, IRCCS San Raffaele
Other Study IDs: 3DD
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Neoplasms; Distal Pancreatectomy (DP)
Keywords: pancreatic disease; early discharge
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases | interventions — Drainage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surgical cohort: All adult patients undergoing elective minimally invasive distal pancreatectomy
  Interventions: Procedure: 3 days discharge

INTERVENTIONS:
Procedure: 3 days discharge — Patients scheduled for elective minimally invasive DP, eligible for the study and willing to participate will be asked to sign the consent form in person during the preoperative counseling session.
  Participants will receive comprehensive preoperative education and will be enrolled in an ERAS protocol that includes urinary catheter removal, initiation of a solid food diet, cessation of intravenous infusions, and oral pain management starting on postoperative day (POD 1). Following discharge on POD3, patients will receive a daily telephonic follow-up by a nurse navigator for the first 7 days after surgery (POD 7).

SUMMARY:
Background: Enhanced recovery after surgery (ERAS) programs and the minimally invasive approach have significantly improved recovery outcomes following distal pancreatectomy (DP). Nevertheless, most patients stay in the hospital a median of 7 postoperative days after laparoscopic DP, despite achieving functional recovery 3-4 days earlier. Early discharge protocols have proven to be safe and feasible If selected patients.

Research objectives: This study aims to evaluate the feasibility and effectiveness of a three-day discharge (3DD) protocol for patients undergoing minimally invasive DP.

Study design: This is an observational, prospective cohort study that will be conducted at San Raffaele Hospital (Milan, Italy) Primary Objective: To investigate the feasibility of a 3-day discharge protocol following a minimally invasive distal pancreatectomy, with post-discharge phone follow-up conducted by a nurse navigator.

Secondary Objective: To investigate the effectiveness of a 3-day discharge protocol following a minimally invasive distal pancreatectomy, evaluate the rate of 30-day emergency departement visits, hospital readmission and patient satisfaction Population: All adult patients undergoing elective minimally invasive distal pancreatectomy who meet the following inclusion criteria will be included in this study

* adult (age>= 18 years) patients undergoing elective minimally invasive distal pancreatectomy
* patients residing or with a temporary accommodation within 50 km or a 30-minute drive from the hospital;
* patients with an adequate support system at home (defined as 24-hour support for at least the first POD7);
* no contraindications to intrathecal or opioid-sparing analgesia;
* patient who have signed the inform consent for participation in the trail;
* No preoperative medical issue requiring inhospital observation longer than three days Patients scheduled for elective minimally invasive DP, eligible for the study and willing to participate will be asked to sign the consent form in person during the preoperative counseling session.

Participants will receive comprehensive preoperative education and will be enrolled in an ERAS protocol that includes urinary catheter removal, initiation of a solid food diet, cessation of intravenous infusions, and oral pain management starting on postoperative day (POD 1). Following discharge on POD3, patients will receive a daily telephonic follow-up by a nurse navigator for the first 7 days after surgery (POD 7).

Preoperatively: patients will complete in person during the counseling visit Patient-Reported Outcomes Measurement Information System (PROMIS)-29 questionnaire and patient-activation measure (PAM) - 13 questionnaires.

At discharge: patients will complete in person in the department PROMIS-29 questionnaire.

At 30 days after surgery, patients satisfaction will be assessed Duration of subject participation: 6 months Duration of total study period: 18 months

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE Over the years, improvements in the management of patients undergoing pancreatic surgery have contributed to enhancing postoperative outcomes and patient recovery. This progress is largely attributed to the centralization of care in high-volume centers. The integration of minimally invasive techniques (such as laparoscopic and robotic surgery), and the adoption of Enhanced Recovery After Surgery (ERAS) protocols. Despite these advancements, the average length of stay (LOS) after distal pancreatectomy (DP) remains around 5 to 7 days. Extended hospital stays often arise from postoperative complications, which occur in approximately 40% of cases following DP. Among these complications, clinically relevant pancreatic fistula (CR-POPF) is the most frequent, affecting up to one-third of patients. However, in most cases, POPF following DP is managed conservatively by simply maintaining the abdominal drain placed intraoperatively. POPF can eventually lead to intra-abdominal fluid collections but rarely to more severe complications such as delayed gastric emptying (DGE), and post-pancrectomy hemorrhage (PPH). Delays in hospital discharge often occur in patients who have already achieved functional recovery, but stay in the hospital due to nonclinical factors such as healthcare system culture or concerns from both surgeons and patients about early discharge.

An early discharge program in selected patients has been successfully demonstrated in colorectal and bariatric surgery. Studies indicate that performing these procedures in an outpatient setting is both feasible and safe, provided upon careful patient selection, patient education, strict adherence to ERAS protocols, and effective follow-up via phone or app-based systems. The advantages of outpatient surgery have been shown to reduce healthcare costs and decrease the wait times for surgery while maintaining equivalent care quality and readmission risk. Although outpatient surgery would be unrealistic for pancreatic surgery, an early discharge program (i.e., before POD5) to patients undergoing DP could yield similar benefits as observed after colorectal surgery. However, the feasibility of an early discharge program has yet to be evaluated in this specific population. The hypothesis is that an early discharge protocol could be effective and feasible in patients undergoing minimally invasive DP, within a preoperative educational program and an adequate telephone follow-up after discharge, without increasing access to ED visits or hospital readmission.

Previous experience and ongoing studies The Division of Pancreatic Surgery at San Raffaele Hospital is among the leading centers for pancreatic surgery in Italy, performing over 300 pancreatic resections annually for the past five years. A prospective quality-improvement registry has been maintained since 2015, encompassing perioperative data from over 2000 patients. In 2023 alone, our division conducted 340 pancreatic resections, including 205 pancreatoduodenectomies, 106 distal pancreatectomies, and 23 total pancreatectomies.

For DP, a minimally invasive approach is preferred for patients with benign or selected malignant lesions, based on factors such as lesion location, vascular involvement, and extent of parenchymal resection required. In our experience, approximately two-thirds of DPs are performed laparoscopically, with a conversion rate to open surgery lower than 10%. Postoperative discharge typically occurs around 7 days after surgery (IQR 6-10), with functional recovery achieved by day 5 (IQR 4-6). Discharge criteria include the ability to tolerate solid food, independence from intravenous fluids, restored gastrointestinal function, sufficient pain management with oral analgesics, independent mobilization, the absence of clinical complications, and the patient's willingness to leave the hospital. In our previous experience, 30% of patients achieved discharge criteria within three days after surgery and underwent an early discharge without 30-day emergency department (ED) visits or hospital readmission, underling the safety of an early discharge protocol. Similar results were found in a different study by the University Hospital Southampton researchers, where they have shown that implementation of ERP (enhanced recovery programme) optimizes outcomes for laparoscopic distal pancreatectomy, with significant earlier return to normal gut function and reduced length of stay, with a median length of stay of 3 days after surgery, without increasing the readmission rate.

For patients with pancreatic fistula, discharge often involves an abdominal drain, with follow-up outpatient visits on POD 7 and POD 15.

Our previous studies show that 19% of patients undergoing laparoscopic DP require emergency department visits (ED) after discharge, and 76% of these patients are readmitted to the hospital, primarily due to intra-abdominal collections. Currently, around 25% of patients are discharged with an abdominal drain due to the presence of an amylase-rich fluid in the abdominal drain. However, previous studies have shown that keeping the drain in place for elevated postoperative amylase levels does not significantly protect against intra-abdominal collections, which may still require antibiotics or operative management. Additionally, the median time for hospital readmission is three weeks after surgery and most postoperative CT scans that reveal complications are performed beyond 10 days after surgery, suggesting that a short hospital stay would not impact readmission rates or necessitate additional interventions. Considering these factors and the PANDORINA trial which underlines the feasibility and safety of a no-drain policy after DP with a reduction in CR-POPF and length of stay, a no-drain approach for patients undergoing minimally invasive DP is adopted. In cases of intraoperative complications or when deemed necessary by the surgeon, an abdominal drain is placed with amylase levels measured on POD1 and POD3. Drains are removed on POD1 if amylase levels are <2000 U/L.

Research Objective:

The objective of this study is to investigate the feasibility and effectiveness of a 3-day discharge protocol following a minimally invasive distal pancreatectomy, with post-discharge phone follow-up conducted by a nurse navigator, which is a nurse uniquely qualified to provide phone support to patients and caregivers throughout the care trajectory and to collect information about clinical health conditions of patients after surgery,

Research Hypothesis:

Our observational prospective cohort study is designed to address several key research questions:

* Can patients undergoing minimally invasive distal pancreatectomy be feasibly discharged on POD3?
* Is POD3 discharge effective for patients following minimally invasive distal pancreatectomy?
* What is the rate of 30-day emergency department visits and hospital readmissions associated with an early discharge protocol?
* What are the primary reasons for emergency department visits, and which of these are potentially preventable?
* How satisfied are patients with the early discharge protocol?

OBJECTIVES AND ENDPOINTS Primary Objective: To investigate the feasibility of a 3-day discharge protocol following a minimally invasive distal pancreatectomy, with post-discharge phone follow-up conducted by a nurse navigator.

Secondary Objective: To investigate the effectiveness of a 3-day discharge protocol following a minimally invasive distal pancreatectomy, evaluate the rate of 30-day emergency departement visits, hospital readmission and patient satisfaction Primary Outcome The feasibility of the 3DD protocol, will be defined as successful discharge on Post Operative Day (POD)3 without any Emergency Department (ED) visits within POD7. The benchmark for feasibility will be considered at 75% Secondary Outcome Effectiveness defined as no development of severe complications (Clavien Dindo Classification ≥ 3) within 7 POD.

STUDY DESIGN This is an observational prospective cohort study that will be conducted at San Raffaele Hospital (Milan, Italy) and was developed according to STROBE guidelines

Study duration Duration of enrollment: 12 months Duration of total follow-up: 6 months Duration of total study period: 18 months

In the Division of Pancreatic Surgery, approximately 110 patients undergo DP each year and 70 are performed laparoscopically. Considering a similar 43% preoperative exclusion rate and a potential 23% dropout rate post-enrollment reported in previous colorectal population, the estimated recruitment period to achieve the target sample size of 30 patients is approximately 12 months. With an additional 6 months required to finalize patient follow-up, data analyses, and manuscript preparation. The time required to complete this study is approximately 18 months.

STUDY POPULATION All patients undergoing elective minimally invasive distal pancreatectomy who meet the following inclusion criteria will be included in this study.

Inclusion Criteria

* adult (age≥ 18 years) patients undergoing elective minimally invasive distal pancreatectomy
* patients residing or with a temporary accommodation within 50 km or a 30-minute drive from the hospital;
* patients with an adequate support system at home (defined as 24-hour support for at least the first POD7);
* no contraindications to intrathecal or opioid-sparing analgesia;
* patients who have signed the informed consent for participation in the trial;
* no preoperative medical issue requiring inhospital observation longer than three days Exclusion Criteria
* Patients undergoing multi-visceral resection;
* undergoing an open procedure;
* requiring vascular resection;
* having a history of chronic opioid use;
* having significant comorbidities or an American Society of Anesthesiologists (ASA) score > 3;
* patients unable to speak Italian;
* having a cognitive impairment;
* developing intraoperative complications; difficulty to be reached after discharge (e.g., limited access to a telephone).

STUDY OBJECT This study aims to evaluate the feasibility and safety of a three-day discharge (3DD) protocol for patients undergoing minimally invasive DP. All procedures, clinical evaluations and follow-up will correspond to current clinical practice.

Study object description Preoperative counseling During preoperative counseling with a surgical resident, all patients will receive information about the surgical procedure, expected postoperative care, and scheduled follow-up after discharge, both verbally and through informational booklets Intraoperative anesthesia and procedure The anesthetic regimen will adhere to institutional guidelines (see Appendix 2). Prior to the surgical procedure, all patients will receive intrathecal analgesia with morphine administered at the T7-9 level (0.15-0.2 ml). General anesthesia will be induced with fentanyl (1-2 mcg/kg), propofol (2 mg/kg), and either rocuronium (0.6 mg/kg) or cisatracurium (0.5 mg/kg), with maintenance provided by inhaled anesthetics.

Surgical procedure: all patients will undergo elective minimally invasive distal pancreatectomy with or without splenectomy. A Pfannenstiel incision will be used for specimen extraction. In patients deemed at high risk of pancreatic fistula according to validated risk scores (e.g., Distal Fistula Risk Score) or experiencing intraoperative complications, the placement of an abdominal drain at the end of the surgical procedure will be considered. In all other patients, no abdominal drain will be placed.

In-hospital postoperative care Postoperative analgesia will be managed with acetaminophen administered three times a day around the clock, along with NSAIDs as needed, starting at the end of surgery. On POD 1, oral tapentadol will be initiated at a starting dose of 50 mg every 12 hours, with this therapy discontinued after POD 7. A detailed ERAS protocol can be found in Appendix 2.

On POD 0, all patients will begin oral fluid intake 6 hours post-surgery, along with intravenous crystalloid infusion at a rate of 2 ml/kg/h.

On POD 1, the urinary catheter will be removed, intravenous infusion will be discontinued, and a solid diet will be introduced. A nurse or physiotherapist will assist with patient mobilization for 30 minutes, twice a day. Patients who tolerate a solid diet without nausea or vomiting, achieve adequate pain control with oral analgesics (NRS ≤ 3 at rest or ≤ 5 during movement), and demonstrate independent mobilization, without complications on POD 2 will be eligible for discharge on POD 3.

Amylase levels will be measured on POD 1 and 3 in patients with an abdominal drain. If the amylase level is less than 2000 U/L on POD 1, the drain will be removed; otherwise, it will remain in place until POD 3. If the amylase level on POD 3 exceeds three times the normal serous value, the patient will be discharged with the drain; if not, the drain will be removed prior to discharge.

Discharge POD 3 Patients who, according to clinical practice, are considered dischargeable on the 3rd day after surgery, are those who meet the following discharge criteria: the ability to tolerate solid food, independence from intravenous fluids, restored gastrointestinal function, sufficient pain management with oral analgesics, independent mobilization, the absence of clinical complications, and the patient's willingness to leave the hospital. In addition, residence or temporary accommodation within 50 km or a 30-minute drive from the hospital, availability of an adequate home support system (defined as 24-hour assistance for at least the first 7 postoperative days) and the opportunity to be reachable by phone upon discharge

At-home postoperative follow-up The nurse navigator will contact the patient daily from POD4 to POD7 to gather information about blood pressure, heart rate, resting saturation, body temperature, diuresis, bowel movements, and the ability to drink or eat. In the presence of an abdominal drain, information will be collected regarding the appearance and 24-hour output, as well as pain assessment. Regarding the last issue, patients will be asked to rate their pain by choosing a number that best represent their current level of pain using a numerical rating scale (NRS) from 0=no pain to 10= worst imaginable pain. A sufficient pain management is considered < 5 (moderate pain) . In case any issues arise after the patient has been discharged and is at home, there is always a ward phone number available, the number of the nurses' station, which is operational 24/7 and can be contacted by the patient at any time.

Preoperatively, patients will complete in person during the counseling visit Patient-Reported Outcomes Measurement Information System (PROMIS)-29 questionnaire and patient-activation measure (PAM) - 13 questionnaires. If patients will be discharged on POD3, they will complete in person in the department PROMIS-29 questionnaire. In case of delayed discharge than POD3, dropping out from the study, the surgeon will complete an interview about the medical reasons and concerns. At 30 days after surgery, patient satisfaction will be assessed using a 5-level Likert scale. Figure 1 provides a detailed overview of the assessment timepoints and corresponding data collection.Figure 1. Data collection at each time point Potential Pitfalls The main potential pitfalls of this observational prospective cohort study may lie in patient enrollment. In previous studies on same-day discharge protocols for colorectal surgery, 43% of candidates were excluded during screening, primarily due to living more than 50 km from the hospital or lacking adequate home support. Among those who met eligibility criteria, an additional 23% were ultimately not discharged as planned due to intraoperative complications, patient refusal, or other medical concerns. In our population, around 40% of patients live in other regions of Italy and would require more than 30 minutes of travel to reach San Raffaele Hospital in Milan, limiting their eligibility. However, many patients with their caregivers find accommodations very close to the hospital during the perioperative, which could increase the number of patients eligible for this study.

Moreover, adherence to the three-day discharge protocol may vary, as surgeons could be hesitant to discharge patients on day three based on individual clinical assessments, particularly if recovery progress is uncertain. Additionally, patients may decline discharge on POD3, especially if a drain is still in place. Previous studies on early discharge programs were largely conducted during the COVID-19 pandemic, a period that heightened patients' motivation to minimize hospital stays due to exposure risks. Without this external motivator, there will be possible enrollment challenges, as patients may be less inclined to embrace a shorter hospital stay.

Subject Recruitment and Screening Pancreatic surgeons will identify potential participants at the outpatient clinic. Eligible patients scheduled for elective minimally invasive DP will be informed about the study by their primary surgeon during the preoperative consultation. Those who express interest will be advised that a member of the study team will contact them to discuss the study in detail during their next visit to the preoperative assessment clinic or by telephone. Additionally, the surgeon will notify the study coordinator about the patient's interest in the study. Patients who are eligible and willing to participate will be asked to sign the consent form in person during the preoperative counseling session.

Subject Identification Starting from the signature of the informed consent by the patient or patient's legal tutor, the subjects is considered enrolled in the clinical study.

A subject identification code will be assigned consecutively. A patient identification list will be kept.

Baseline Assessments Pancreatic surgeons will identify potential participants at the outpatient clinic. (1) Eligible patients scheduled for elective minimally invasive DP will be informed about the study by their primary surgeon during the preoperative consultation. (2) Those who express interest will be advised that a member of the study team will contact them to discuss the study in detail during their next visit to the preoperative assessment clinic or by telephone. Additionally, the surgeon will notify the study coordinator about the patient's interest in the study. (3) Patients who are eligible and willing to participate will be asked to sign the consent form in person during the preoperative counseling session.

Preoperatively, patients will complete in person during the counseling visit Patient-Reported Outcomes Measurement Information System (PROMIS)-29 questionnaire and patient-activation measure (PAM).

Visits and Follow Up The nurse navigator will contact the patient daily from POD4 to POD7 to gather information about body temperature, diuresis, bowel movements, and the ability to drink or eat. In the presence of an abdominal drain, information will be collected regarding the appearance and 24-hour output, as well as pain assessment using a numerical rating scale (NRS). A phone number and an email address will be provided for clinical questions or concerns from 7:00 a.m. to 5:00 p.m., 5 days per week. Outside of working hours, patients will be informed about the option to present to go to the emergency room. Patients without postoperative drains will undergo a follow-up in outpatient setting at 15 and 30 days after surgery. In case of drain after discharge additional follow-up will be conducted weekly until drain removal.

Definition of End of Study According to the study design, the end of the study is defined as the date on which the last patient completes the last visit: 30 days after surgery

Premature termination or suspension of a study This study may be temporarily suspended or prematurely terminated by the authorized Sponsor representative or the PI if there is sufficient reasonable cause related to investigators decisions

DATA MANAGEMENT Definition of source data and source documents Source data are contained in source documents (original records or certified copies). Any data recorded directly on the CRFs (i.e., no prior written or electronic record of data), is considered to be source data.

Source Documents: Original documents, data, and records (e.g., hospital records; clinical and office charts; laboratory notes; memoranda; subjects' diaries or evaluation checklists; pharmacy dispensing records; recorded data from automated instruments; copies or transcriptions certified after verification as being accurate copies, microfiches, photographic negatives, microfilm or magnetic media, x-rays, subject files, or records kept at the pharmacy, at the laboratories, and at medico-technical departments involved in the clinical study).

All parameters asked for in the case report form (CRF) will be documented in the source documents.

A record of patient screen failures will be maintained for patients who do not qualify for enrollment, including the reason for the screen failure.

Documentation of data in Case Report Forms (CRFs) All relevant data collected during the study for all patients enrolled in the study will be collected in the eCRF (RedCAp) by the investigator responsible or someone authorized by the investigator in a timely manner (as soon as possible after the information is collected) to ensure that it is clear and legible. The physician must confirm the completeness, correctness, plausibility and compliance with ICH guidelines and institutional SOPs of the data by dated signature. An explanation must be provided for any and all missing data.

REDcap is a clinical electronic data capture system specifically developed around HIPAA-Security guidelines; more information on the consortium and system security is available at https.//www.projectredcap.org/.

A copy of all pages will be conserved in the study site.

Data Protection

The Investigator undertakes to:

* use the data only for the purposes of the foreseen analyses and within the limits established by the study and approved by the competent EC;
* store data in a secure network system;
* prohibit unauthorised third parties from accessing, even partially, data.
* guarantees to limit access to and processing of data only to its employees and collaborators who, upon appointment as an authorized person:

  1. need to process the data in order to carry out their work in relation to the study;
  2. have undertaken to maintain the confidentiality of the Data and of any information deriving from it or that is communicated to them.

If, within the context of the Study, the Investigator needs to make use of its own suppliers, the latter undertakes to appoint these subjects as Data Processors /Responsabili dei Trattamenti with a specific agreement or other legal act suitable for this, before the start of any data processing by them, according to Regulation (EU) n. 2016/679, art. 28.

The Investigator also undertakes to adopt suitable measures to facilitate the exercise of the rights of the subject provided for by Regulation (EU) n. 2016/679, art. 15 - 22, including the rights of access, rectification, cancellation, limitation, opposition and portability, within 30 days of receiving the relative request.

In case the Investigator need to communicate the data outside OSR (the Data Controller /Titolare) in pseudonymized form, the Investigator will refrain from carrying out any activity aimed at identifying the identity of the subjects to whom such data refer.

STATISTICS Description of Statistical Methods Categorical variables will be presented as counts and percentages, while continuous variables will be reported as means with standard deviations (SD) or as medians with interquartile ranges (IQR), as appropriate.

Sample Size Determination The feasibility of the 3DD protocol, has be defined as successful discharge on POD 3 without any ED visits within POD7. Our previous studies show that 19% of patients undergoing laparoscopic DP require emergency department visits (ED) after discharge, and 76% of these patients are readmitted to the hospital, primarily due to intra-abdominal collections. Therefore it is defined a benchmark of 75% to stay under the standard of care.

To estimate a success rate of successful discharge on POD 3 of 75%, with a margin of error of 10% and a confidence level between 80 and 85%, a minimum of 35 patients is required.

Statistical Design To assess the feasibility of 3DD with a target success rate of at least 70%, a sample size of 30 patients is deemed sufficient. Categorical variables will be presented as counts and percentages, while continuous variables will be reported as means with standard deviations (SD) or as medians with interquartile ranges (IQR), as appropriate. Subgroup analyses will compare patients discharged with a drain versus those discharged without one.

ELIGIBILITY:
Inclusion Criteria:

* adult (age>= 18 years) patients undergoing elective minimally invasive distal pancreatectomy
* patients residing or with a temporary accommodation within 50 km or a 30-minute drive from the hospital;
* patients with an adequate support system at home (defined as 24-hour support for at least the first POD7);
* no contraindications to intrathecal or opioid-sparing analgesia;
* patient who have signed the inform consent for participation in the trail;
* No preoperative medical issue requiring inhospital observation longer than three days

Exclusion Criteria:

* Patients undergoing multi-visceral resection;
* undergoing an open procedure;
* requiring vascular resection;
* having a history of chronic opioid use;
* having significant comorbidities or an American Society of Anesthesiologists (ASA) score > 3;
* patients unabled to speak Italian;
* having a cognitive impairment;
* develoing intraoperative complications;
* difficulty to be reached after discharge (e.g., limited access to a telephone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing elective minimally invasive distal pancreatectomy who meet the following inclusion criteria will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-09-13 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients without any Emergency Department (ED) visits within POD7 | 7 days after surgery
  The feasibility of the 3DD protocol, will be defined as successful discharge on Post Operative Day (POD)3 without any Emergency Department (ED) visits within POD7. The benchmark will be considered at 75%.

SECONDARY OUTCOMES:
Percentage of patients with no development of severe complications within 7 POD | 7 days post surgery and 30 days post surgery
  Effectiveness of early discharge is defined as no development of severe complications (Clavien Dindo Classification ≥ 3) within 7 POD.